CLINICAL TRIAL: NCT05615064
Title: Evaluation of the Relationship Between Quality of Life, Life Satisfaction and Anxiety Levels of Wheelchair Basketball Players
Brief Title: Relationship Between Quality of Life, Life Satisfaction and Anxiety Levels of Wheelchair Basketball Players
Status: Completed | Type: Observational
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Other Study IDs: 202206Y0254
Record Dates: First submitted 2022-11-02; First posted 2022-11-14 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Quality of Life; Life Satisfaction; Anxiety Levels
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: relationship between quality of life, life satisfaction and anxiety levels of wheelchair basketball players — relationship between quality of life, life satisfaction and anxiety levels of wheelchair basketball players

SUMMARY:
Today, there are many studies on wheelchair basketball players. However, these studies do not indicate the relationship between the quality of life, life satisfaction and anxiety levels of wheelchair basketball players, in the extent of the knowledge. As a result of this study, it is aimed to obtain information about the quality of life, life satisfaction and anxiety levels of wheelchair basketball players.

DETAILED DESCRIPTION:
The study aimed to examine the relationship between the quality of life, life satisfaction and anxiety levels of wheelchair basketball players. This study was carried out with wheelchair basketball players in Istanbul between March 2022 and May 2022. Twenty-three wheelchair basketball players were included in the study. The scope of the study was explained to the wheelchair basketball players who participated in the study during the face-to-face interview, and the consent forms prepared by the researcher were distributed. The participants, who approved the consent form and agreed to participate in the study, had to fill out the sociodemographic form. The quality of life of the participants was determined by the SF-12 Quality of Life Scale; Satisfaction with life was evaluated with the Satisfaction with Life Scale, and anxiety levels were evaluated with the Beck Anxiety Scale. Statistics were performed using SPSS Version 22.0 program.

ELIGIBILITY:
Inclusion Criteria:

* Being between the age of 18-45
* Participating in a wheelchair basketball team regularly
* Being disabled regardless of the disability score

Exclusion Criteria:

● Being over the age of 45

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: wheelchair basketball players
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2022-11-06 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-26 (Actual)

PRIMARY OUTCOMES:
Sociodemographic Features | 3 weeks
  The question include the participants age, gender, education level, years of experience
Assesment of Quality of Life | 3 weeks
  SF-12 is the short form of the SF-36 which is a gold standart used to asses quality of life in individuals. The questionnaire is also reported either physical (SF12-PCS) or mental component summary scale (SF12-MCS), the regression weightings used for scoring the SF12 come from a general population.
Assessment of Life Satisfaction | 3 weeks
  The Satisfaction With Life Scale (SWLS) was developed to assess satisfaction with the respondent's life as a whole. It consists of 5 items with one dimensional structure and it's rated from 1(completely disagree) to 5 (completely agree)
Assessment of Anxiety | 3 weeks
  The BAI is a 21-items self-report questionnaire that lists symptoms of anxiety. A total score for the BAI is obtained by summing the ratings of the 21-items.

CONTACTS AND LOCATIONS:
Locations (1):
- Yeditepe University, Istanbul, Turkiye, Turkey (Türkiye)